CLINICAL TRIAL: NCT02290418
Title: Prospective Randomized Controlled Clinical Study Comparing Two Bariatric Bypass Procedures, Roux-en-Y Gastric Bypass (RYGB) and Omega-Loop Gastric Bypass (OLGB), in Patients With Severe Obesity and Metabolic Disease
Brief Title: Roux-en-Y Gastric Bypass (RYGB) Versus Omega-Loop Gastric Bypass (OLGB) Safety and Efficacy Short-term Study
Acronym: ROSESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nemocnice Břeclav, p.o. (Other)
Responsible Party: Principal Investigator, Dr. Michal Cierny, PhD, bariatric surgeon, Nemocnice Břeclav, p.o.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYGBvsOLGB
Record Dates: First submitted 2014-10-31; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Obesity, Severe; Diabetes Mellitus, Type 2
Keywords: Roux-en-Y Gastric Bypass; Omega-Loop Gastric Bypass; "Mini-Gastric" Bypass
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y Gastric Bypass (Active Comparator): Laparoscopic Roux-en-Y Gastric Bypass and routine care.
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Omega-Loop Gastric Bypass (Active Comparator): Laparoscopic Omega-Loop Gastric Bypass and routine care.
  Interventions: Procedure: Omega-Loop Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — Laparoscopic Gastric Bypass performed with two anastomoses (gastro-enteral and entero- enteral), two limbs (Alimentary limb of length 150cm and Biliary limb of length 75-100cm) and sewing of mesenteric defect.
  Other Names: RYGB
  Arms: Roux-en-Y Gastric Bypass
Procedure: Omega-Loop Gastric Bypass — Laparoscopic Gastric Bypass performed with single anastomosis (gastro-enteral) connecting a long gastric pouch to small bowel with Afferent limb of length 200cm.
  Other Names: OLGB; Mini-Gastric Bypass; Single Anastomosis Gastric Bypass
  Arms: Omega-Loop Gastric Bypass

SUMMARY:
The aim of this study is to compare the relative clinical outcomes between two variants of gastric bypass [Roux-en-Y Gastric Bypass (RYGB) or Omega-Loop Gastric Bypass (OLGB)] in metabolic surgery candidates with Body Mass Index (BMI) between 35 and 50. The study will examine the short and medium term effects of each intervention on weight, obesity comorbidities, quality of life and gastroscopy findings.

DETAILED DESCRIPTION:
Introduction:

Obesity is a risk factor for Diabetes, Ischemic heart disease, Stroke, and Hypertensive heart disease, which are the 6th, 1st, 2nd, and 10th leading causes of death according to the WHO. Bariatric or Metabolic Surgery is an Efficient and reasonably Safe method for the Treatment of Severe Obesity, Type 2 Diabetes (T2DM) and Metabolic Syndrome (MS).

Existing knowledge:

Metabolic procedures, e.g. Gastric bypass, are more effective in the treatment of T2DM than predominantly "restrictive" procedures, e.g. Gastric Banding. RYGB is one of the most prevalent procedures in the world and Europe. In the USA, RYGB is considered a "golden standard" in bariatric surgery. In the recent decade, a simpler variant of Gastric bypass, i.e. OLGB, has been proposed. Proponents of OLGB argue it has less complications and seems to have higher and more durable effect on weight reduction and T2DM improvement. Opponents of OLGB are concerned that chronic exposure of gastric or esophageal mucosa to bile, as seen in animal experiments and in patients operated for gastric cancer or peptic ulcer disease, pose a severe health risk. So far, this concerns has not been confirmed in OLGB patients. Only one Randomized Controlled Trial (RCT) of these two interventions was performed, concluding OLGB to be simpler and safer with a similar Efficacy 2 years after the surgery.

Need for a trial:

A growing evidence supports the efficacy and safety of bariatric and metabolic surgery for the treatment of severe obesity and T2DM. Therefore, bariatric surgery is being more frequently performed. However, there is little evidence from randomized trials comparing different bariatric procedures - most comes from retrospective cohorts, which might suffer from bias. As a result, the choice of a bariatric procedure for a particular patient is based largely on the preference and experience of the particular surgeon, rather than evidence of best benefit for a particular patient. Although the efficacy and safety of RYGB is well established, newer variants or other less frequently employed bariatric procedures might offer more preferable Efficacy or Safety profile for some patients. Some evidence suggests OLGB might a promising procedure, which is "simpler and safer with similar efficacy" in comparison to RYGB, a technically more demanding procedure. This study contributes with rigorous evidence to further define the relative strengths and weaknesses of OLGB as compared to the "gold standard" RYGB.

Objectives:

The purpose of this study is to objectively compare the efficacy of RYGB and OLGB on weight, T2DM and other obesity-related comorbidities. Furthermore, this study aims to provide more insight into the safety of OLGB and RYGB by measuring the incidence of complications and abnormal findings on Gastroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Severe Obesity: BMI ≥ 40 and ≤ 50 or (BMI ≥ 35 and < 40 and type 2 diabetes or metabolic syndrome)
* Inadequate results of Attempts to loose weight by Conservative means
* Ability to understand the nature of the procedure and willing to follow postoperative routine lifestyle and checkups
* no contraindication for bariatric surgery on psychological assessment
* no contraindication for general anesthesia
* consent for both variants of gastric bypass surgery
* consent to participate in a study with randomized design

Exclusion Criteria:

* prior bariatric surgery of any kind
* gravidity or recent (<1 year) labour
* drug or alcohol abuse
* symptomatic Gastro Esophageal Reflux Disease (GERD)
* hiatal hernia, > 3cm
* esophagitis, ≥ 2. grade
* active smoker
* chronic renal disease, stage ≥ 3
* patient immobility
* surgery not covered by universal insurance in Czech rep. (i.e. international patients)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite measure of success of bariatric surgery as measured by Bariatric Analysis and Reporting Outcome System (BAROS) | baseline, 1 and 2 years
  BAROS composite score rates weight loss, change in comorbidities, and quality of life.

SECONDARY OUTCOMES:
Change in weight, measured as Percent of Excess Weight Loss (%EWL) | baseline, 1 and 2 years
Change in weight, measured as Percent of Excess Body Mass Index Loss (%EBMIL) | baseline, 1 and 2 years
Change in Type 2 Diabetes Mellitus, measured as intensity of medical treatment: increased, same, decreased, or discontinued | baseline, 1 and 2 years
Change in Type 2 Diabetes Mellitus, measured as intensity of treatment: diet alone, oral antidiabetic agent(s), insulin (IU/day) | baseline, 1 and 2 years
Durability of change in Type 2 Diabetes Mellitus, measured as proportion of patients with T2DM partial remission who experience T2DM "relapse" | 2 years
Change in Hypertension, measured as intensity of medical treatment: increased, same, decreased, or discontinued | baseline, 1 and 2 years
Change in Dyslipidemia, measured as intensity of medical treatment: increased, same, decreased, or discontinued | baseline, 1 and 2 years
Change in Obstructive Sleep Apnea (OSA), measured as the need of use of mouth device | baseline, 1 and 2 years
Change in Obstructive Sleep Apnea, measured as score on Epworth questionnaire scale | baseline, 1 and 2 years
Incidence of Ulcer or other Abnormal Finding on Endoscopic Gastroscopy, measured as proportion of patients with abnormal finding in each arm | 1 and 2 years
Incidence of Ulcer or other Abnormal Finding on Endoscopic Gastroscopy, measured as Rate of unique Event per 100 patient-years of follow up | up to 5 years
Incidence of early postoperative (<=30 days) Reoperations and Complications of grade >= 2 according to Clavien-Dindo classification | 30 days
Incidence of late (>30 days) Reoperations, Complications, and detected adverse outcomes | 1 and 2 years
Incidence of Reoperations, Complications, and detected adverse outcomes, measured as Rate of Event per 100 patient-years of follow up | up to 5 years
Change in Quality of Life, as measured by Moorehead-Ardelt Questionnaire II | baseline, 1 and 2 years

OTHER OUTCOMES:
Operative time, measured in minutes | intraoperative
Length of inpatient stay due to performance of assigned intervention, measured in days | recorded at time of discharge, estimated average 4 days from the surgery
  number of days from the day of surgery (Post Operative Day 0) until the end of hospitalization
Change in body weight, measured as proportion of patients with EWL > 50%, and proportion of patients with EWL < 25% | baseline, 1 and 2 years
Change in body weight, measured in kilograms (kg) | baseline, 1 and 2 years
Change in Body Mass Index (BMI), measured in kg/m2 | baseline, 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michal Cierny, Dr., Study Director — Breclav Hospital
Locations (1):
- Bariatric Clinic, Breclav Hospital, Břeclav, Czechia

REFERENCES:
- See also: Laparoscopic Roux-en-Y versus mini-gastric bypass for the treatment of morbid obesity: a prospective randomized controlled clinical trial. — http://www.ncbi.nlm.nih.gov/pubmed/15973097?dopt=Abstract
- See also: Laparoscopic Roux-en-Y Vs. Mini-gastric Bypass for the Treatment of Morbid Obesity: a 10-Year Experience — http://link.springer.com/article/10.1007/s11695-012-0726-9
- See also: Greater Weight Loss with the Omega Loop Bypass Compared to the Roux-en-Y Gastric Bypass: a Comparative Study — http://link.springer.com/article/10.1007/s11695-014-1180-7
- See also: "Mini" Gastric Bypass: Systematic Review of a Controversial Procedure — http://link.springer.com/article/10.1007/s11695-013-1026-8
- See also: Weight Loss Surgery Results — http://wlsr.eu
- See also: Interdisciplinary European guidelines on metabolic and bariatric surgery. — http://www.ncbi.nlm.nih.gov/pubmed/24081459